CLINICAL TRIAL: NCT02080663
Title: Long-term Outcome of Proximal Row Carpectomy. Influence of the Shape of the Capitate
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Pellenberg (Other)
Responsible Party: Principal Investigator, Maarten Van Nuffel, Fellow Upper Limb Surgery, University Hospital Pellenberg
Other Study IDs: PRC Van Nuffel De Smet
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Wrist Arthritis
Keywords: carpectomy, proximal row, long-term, wrist, arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Proximal row carpectomy: Proximal row carpectomy
  Interventions: Procedure: Proximal row carpectomy

INTERVENTIONS:
Procedure: Proximal row carpectomy

SUMMARY:
In cases of severe arthritis of the wrist, surgical removal of the scaphoid, lunate and triquetrum bones or proximal row carpectomy (PRC) is a well-known procedure. This procedure converts the wrist in a simple hinged joint but allows us to preserve a certain range of motion in the wrist. One of the main disadvantages of PRC is the risk of developing arthritis between the head of the capitate and the lunate fossa. The long-term follow-up of this procedure has always been a reason for concern. The investigators set up this retrospective study to evaluate the long-term results of the procedure in the investigators institution.

Also, the shape of the head of the capitate may play a role in the development of arthritis. A more round shape could distribute the forces more equally and thus prevent the progression of cartilage damage

The study hypothesis is:

* PRC preserves range of motion and force in the long term (more than 10 years postoperatively).
* A more round head of the capitate is associated with an increased risk of developing arthritis in the new joint.

DETAILED DESCRIPTION:
We invite all patients who underwent a PRC at our institution with a follow-up of more than 10 years for review.

Questions

* VAS pain in rest and during activity

  * Pain is quantified as none, minimal (pain with strenuous activity), moderate (pain with daily activity), or severe (pain at rest).
  * If pain, use of analgetics, splint, …
* quick DASH
* patient related wrist evaluation (PRWE) score. form-36 (SF-36) general health status outcome ?
* Satisfaction, do it again?
* Complications? Re-operations?
* Return to work after operation, which job (manual labor?) changed job due to wrist problems? Worker's compensation claims?

Clinical review

* grip force + other side to compare (Jamar Dynamometer)
* pinch grip + other side to compare
* range of motion measurement:

  * absolute and compared to other side
  * flexion-extension, ulnar-radial deviation and prosupination

Radiography:

* Standard anterioposterior and lateral wrist radiography performed to evaluate the onset or degree of arthritis.

  o Radiocapitate arthrosis grading:
  * None
  * Minimal (joint space narrowing alone),
  * Moderate (joint space narrowing with adjacent subchondral sclerosis)
  * severe (bone collapse, erosion, or subchondral cyst formation)
* Oldest radiography of each patient was retrieved and the shape of the capitate evaluated.
* If available, a pre-operative MRI scan could also be interpreted. (Probably no MRI's available, but MRI gives a better indication of the shape of the capitate than plain X-ray).
* Review: documentation of intra-operative findings concerning capitate and lunate fossa.

Statistical analysis

* Student's t-test on the numerical data
* Wilcoxon signed- rank test on the visual analog scales
* Differences significant at p < .05. Two-tailed tests in all cases.
* Subgroups according to initial diagnosis
* Compare results with the initial follow-up to evaluate the prospective value of this follow-up moment.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent a Proximal row carpectomy

Exclusion Criteria:

* Bilateral procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent a Proximal row carpectomy in our institution more than 10 year ago will be contacted for review
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
quick DASH score | more than 10 year after operation
  The Disability of Arm, Shoulder and Hand score is a standardised outcome measure for upper limb evaluation.

SECONDARY OUTCOMES:
Arthritis between capitate and lunate fossa | 10 years after operation
  radiographic evaluation of arthritis in the wrist:
  * None
  * Minimal (joint space narrowing alone),
  * Moderate (joint space narrowing with adjacent subchondral sclerosis)
  * Severe (bone collapse, erosion, or subchondral cyst formation)

OTHER OUTCOMES:
Range of movement | 10 years after operation
  clinical measurement with a goniometer of the flexion, extension, ulnar and radial deviation and pronation and supination + comparison to the other, uninvolved wrist

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Van Nuffel, M.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium